CLINICAL TRIAL: NCT03833882
Title: Evaluation of the Performance of the Tear Substitute MAF-1217 in Patients With Evaporative DED
Brief Title: Evaluation of MAF-1217 in Patients With DED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VF-OS-001/2018
Record Dates: First submitted 2019-01-31; First posted 2019-02-07 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Evaporative Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cationorm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAF1217/Cationorm (Experimental)
  Interventions: Device: MAF1217; Other: Cationorm
- Cationorm/MAF1217 (Experimental)
  Interventions: Device: MAF1217; Other: Cationorm

INTERVENTIONS:
Device: MAF1217 — The study population will have to self-administer the study treatment in a TID posology.
Other: Cationorm — The study population will have to self-administer the study treatment in a TID posology.

SUMMARY:
This is a pre-market, multicentre, double-blind, randomized, crossover, non-inferiority study comparing the efficacy of MAF-1217 and Cationorm® in adult patients with evaporative DED.

The study population will be divided in 4 different subgroups, according to the different types of evaporative DED:

1. Group A: high evaporative levels
2. Group B: females in menopause, whether using hormonal integration or not
3. Group C: presence of active obstructive Meibomian gland disease
4. Group D: glaucomatous patients

DETAILED DESCRIPTION:
Patients will be enrolled after having signed the informed consent form prior any other study procedure and after inclusion/exclusion criteria check.

Each patient will be planned to perform 6 study visits and at each visit all necessary study procedures will be performed according to the clinical investigation plan requirements (see flow-chart).

The study visits will be performed at: screening, baseline, week 2, week 6, week 8, week 12.

Patients will be enrolled at screening visit and at baseline, after the wash-out period of 1 week, then will be randomized to receive MAF-1217 or Cationorm® for the following 6 weeks.

After this time lapse, patients will be switched to the opposite therapy for 6 additional weeks.

The entire study population will be asked for a TID posology, and will be divided in 4 different subgroups, according to the different types of evaporative DED.

Certain test will be performed only in some patients:

Osmolimetry and tear sampling in 20 patients(10/site) chosen random from groups B, C and D; Ferning test only in group D; tear film collection and cytokine expression only in 20 patients form site nr. 2.

Patients will be allowed to carry on any systemic or local medications, apart lubricating eyedrops, which have to be stopped the day before baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old (adult patients), male and female
2. Schirmer I test > 10 mm at 5'
3. (Group A): high evaporative levels
4. (Group B): females in menopause, both using hormonal integration or not
5. (Group C): presence of active obstructive Meibomian gland disease, defined as at least one of the following:

   * Meibomian orifice plugging
   * eyelid margin foaminess
   * changes in orifice position with respect to the mucocutaneous junction
   * abnormal Meibomian gland secretions (opaque and viscous-like form that is difficult to express)
6. (Group D): glaucomatous patients receiving one or more BAK preserved treatments for at least 2 years, showing an abnormal Ferning test (Types 3 or 4 according to Rolando)
7. all: wishing to participate in the study and able to sign the ICF

Inclusion criteria to be checked at baseline:

1. BUT < 7"
2. Mild to severe DED according to OSDI chart

Exclusion Criteria:

1. Neuropathic causes of dry eye (diabetes, long-standing contact lens wearing, previous ocular herpes infections)
2. Coexisting corneal diseases
3. Autoimmune diseases
4. Past or active cicatricial conjunctivitis
5. Past ocular surface burns
6. Keratinization of the eyelid margin
7. Sjogren syndrome
8. History of corneal trauma
9. Pregnant and lactating women
10. Younger than 18 years old patients
11. Use of contact lenses
12. inability to self administer study medications
13. (GROUPS B, D) Presence of active obstructive Meibomian gland disease
14. (GROUP C) Presence of cicatricial Meibomian gland disease
15. known allergic sensitivity to any of the devices ingredients or any other known allergy
16. participation in a clinical trial during the 3 months prior to the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Break-up time (BUT) differences | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Changes in break-up time (BUT) versus baseline

SECONDARY OUTCOMES:
ocular surface staining (corneal and conjunctival) | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Cross-over analysis for the differences versus baseline between the two groups on changes in ocular surface staining (corneal and conjunctival)
Schirmer I test (ST) (without anesthesia) | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Cross-over analysis for the differences versus baseline between the two groups on changes in Schirmer I test (ST) (without anesthesia)
number of blinking per minute | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Cross-over analysis for the differences versus baseline between the two groups on changes in number of blinking per minute
Ferning test (Group D) | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Cross-over analysis for the differences versus baseline between the two groups on changes in Ferning test (Group D)
osmolarity | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Cross-over analysis for the differences versus baseline between the two groups on changes in osmolarity
patient satisfaction (10 points VAS scale) | measured at week 2, 6, 8 and 12 weeks treatment versus baseline
  Cross-over analysis for the differences versus baseline between the two groups on changes in patient satisfaction (10 points VAS scale).
  (VAS: scale where patient has to specify level of satisfaction by indicating a position along a continuous line between two end-points (0 - 10). 0 indicates no satisfaction while 10 represents the highest level).
OSDI | measured at week 2, 6, 8 and 12 weeks treatment
  Changes in questionnaire scores (OSDI - Ocular Surface Disease Index). The overall Ocular Surface Disease score defined the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale San Paolo, ASST Santi Paolo e Carlo, Milan
  - ASST Fatebenefratelli Sacco P.O.L. Sacco, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fogagnolo P, Quisisana C, Caretti A, Marchina D, Dei Cas M, Melardi E, Rossetti L. Efficacy and Safety of VisuEvo(R) and Cationorm(R) for the Treatment of Evaporative and Non-Evaporative Dry Eye Disease: A Multicenter, Double-Blind, Cross-Over, Randomized Clinical Trial. Clin Ophthalmol. 2020 Jun 18;14:1651-1663. doi: 10.2147/OPTH.S258081. eCollection 2020. PMID 32606580